CLINICAL TRIAL: NCT03820869
Title: The Effect Of Occupational Therapy On Sensory-Based Feeding Problems Of Children Wth Autism Spectrum Disorder
Brief Title: The Effect Of Occupational Therapy On Sensory-Based Feeding Problems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özgü İNAL, Assoc Prof, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/454
Record Dates: First submitted 2019-01-18; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Feeding Disorder; Autism Spectrum Disorder; Sensory Integration Disorder (Disorder)
MeSH Terms: conditions — Feeding and Eating Disorders; Autism Spectrum Disorder | interventions — Sex Education; Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Children with ASD
  Interventions: Other: Family Training
- Intervention (Experimental): Children with ASD
  Interventions: Other: Occupational Therapy

INTERVENTIONS:
Other: Family Training — Family Training
  Arms: Control
Other: Occupational Therapy — Occupational Therapy
  Arms: Intervention

SUMMARY:
Feeding problems are common in individuals with Autism Spectrum Disorder (ASD).This study was planned to investigate the effect of occupational theraphy on sensory feeding problems in ASD.

DETAILED DESCRIPTION:
Feeding problems are common in individuals with Autism Spectrum Disorder (ASD).This study was planned to investigate the effect of occupational theraphy on sensory feeding problems in ASD.

ELIGIBILITY:
Inclusion Criteria:

* ASD
* Feeding problems

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Dunn Sensory Profile | 8 weeks
  It is a norm-referenced, parent-report questionnaire. The parent rates frequency of each item on a 5-point Likert scale from 1= always to 5= never. It reports the frequency of behavioural occurrences that are used to measure the patterns of performance indicative of difficulties experienced in sensory processing

SECONDARY OUTCOMES:
BAMBİ | 8 weeks
  The BAMBI is rated based on a parent proxy report, with a 5-point grading type scale (1 = Never/Very Rarely -5 = At Almost All Mealtimes). It was designed to capture mealtime behaviors specific to children with ASD.
STEP | 8 weeks
  It is used for to identify the feeding problems of persons with ID in terms of (a) risk of aspiration, (b) food selectivity, (c) feeding skills deficits, (d) food refusal and associated behavior problems, and (e) nutrition-related behavior problems